CLINICAL TRIAL: NCT06056843
Title: Evaluation of a Handheld Ultrasound Device to Triage Women With a Positive Clinical Breast Examination by Trained Health Workers and Medical Officers
Brief Title: Handheld Ultrasound Device to Triage Women With a Positive Clinical Breast Examination by Trained Non-radiologists
Acronym: PUD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: International Agency for Research on Cancer (Other)
Collaborators: Malabar Cancer Care Society Kannur, India (Unknown); Bhabha Atomic Research Centre (BARC), India (Unknown)
Responsible Party: Principal Investigator, Farida Selmouni, Scientist, International Agency for Research on Cancer
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: IEC 21-04
Record Dates: First submitted 2023-09-21; First posted 2023-09-28 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Breast Cancer; Carcinoma in Situ
Keywords: Breast cancer; Screening; Low- and middle-income countries; Clinical breast examination; Portable ultrasound device; Triage
MeSH Terms: conditions — Breast Neoplasms; Carcinoma in Situ

STUDY DESIGN:
Intervention Model Description: This is a single-arm study in which women with a positive clinical breast examination will be triaged using a portable ultrasound device by non-radiologists. The gold standard is mammography, ultrasound and histology if needed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental): Triage of clinical breast examination positive women using handheld ultrasound by non-radiologists.
  Interventions: Other: Triage of clinical breast examination positive women using handheld ultrasound by non-radiologists.

INTERVENTIONS:
Other: Triage of clinical breast examination positive women using handheld ultrasound by non-radiologists. — Women screened for breast cancer by clinical breast examination (CBE). Those with positive CBE will be triaged by portable ultrasound device by non-radiologists. All recruited women will receive a diagnostic mammography and, if necessary, an ultrasound performed by a radiologist. The radiologist will be blinded to the portable ultrasound device findings. Those with suspected lesions either on mammography or ultrasound will have fine needle aspiration cytology (FNAC) or core biopsy. The women with confirmed diagnosis of breast cancer will be staged and appropriately treated as per the policy of the hospital.

SUMMARY:
Cross sectional study to evaluate estimate accuracy of portable ultrasound device in correctly differentiating the benign breast lesions from the malignant ones in the women referred with a positive Clinical breast examination (CBE) screening test.

DETAILED DESCRIPTION:
More than two million new cases of breast cancer occur each year worldwide. Implementing mammography screening is complex and resource-intensive, making it impractical in resource-limited settings. Clinical breast examination (CBE) has been recommended as an alternative screening option for low- and middle-income countries. Several studies have shown a significant shift towards earlier stage tumours detected by CBE. However, the high false-positive rate and low positive predictive value of CBE expose women to unnecessary and costly further diagnostic procedures, as well as the negative psychological consequences. There is an urgent need for a more accurate, cost-effective and reliable triage technology that can be performed by any healthcare provider.

ELIGIBILITY:
Inclusion Criteria:

* Clinical breast examination positive women with no debilitating illness.
* Symptomatic women found to be positive on clinical breast examination by nurses/midwives or medical officers.

Exclusion Criteria:

* Women with confirmed diagnosis of breast cancer or those already treated for the disease.

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 150 (Estimated)
Dates: Start 2022-05-09 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of non-radiologist portable ultrasound device for triaging women with positive clinical breast examination | Through study completion, an average of 1 year
  Sensitivity, specificity and positive and negative predictive values of portable ultrasound device to detect breast cancer and carcinoma in situ with repeat clinical breast examination, mammography/ultrasound and/or cytology/core biopsy as the gold standard test.

SECONDARY OUTCOMES:
Agreement between portable ultrasound device and mammography/ultrasound | Through study completion, an average of 1 year
  Agreement between portable ultrasound device and mammography/ultrasound by a radiologist in differentiating malignant and benign solid breast lesions.

CONTACTS AND LOCATIONS:
Locations (1):
- Malabar Cancer Care Society Kannur, Kannur, India